CLINICAL TRIAL: NCT00882271
Title: Efficacy of Acupuncture to Improve Symptoms and Functionality for People With Fibromyalgia
Brief Title: Fibromyalgia Acupuncture Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Fibromyalgia Acupuncture Study, Southern California University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCU-08-VINJ003
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Acupuncture; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Traditional Chinese Acupuncture
  Interventions: Other: Acupuncture
- 2 (Placebo Comparator): Placebo Acupuncture
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Ten Acupuncture treatments within six weeks

SUMMARY:
The acupuncture treatment in this study is particularly aimed at reducing the pain and other negative health events such as emotional trauma and disability associated with Fibromyalgia, while improving the quality of life and promoting general health.

DETAILED DESCRIPTION:
It is hypothesized that acupuncture treatment will be effective in reducing pain and improving lower body strength and overall functionality more than the sham acupuncture treatment in people with Fibromyalgia (FM). The purpose of this study is to compare the efficacy of acupuncture with simulated acupuncture in patients with FM using a randomized controlled design. More specifically, the objectives of this study are to determine if acupuncture can (1) reduce pain, (2) improve lower body strength, and (3) improve overall functionality.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older and can be of either sex.
2. A confirmed diagnosis of FM (pain for more than three months) will be required to participate in the study. If they do not have a diagnosis the study clinician or research assistant will examine them and determine their eligibility.
3. All participants must be willing to provide a written informed consent prior to participation and should not have undergone acupuncture treatment in the past.

Exclusion Criteria:

1. Acupuncture treatment in the past five years.
2. Unwilling to sign informed consent.
3. Less than a score of 40 on the Fibromyalgia Impact Questionnaire,
4. Involvement in any litigation currently or in the past,
5. Simultaneous infection with HIV/Hepatitis B virus.
6. Severe depression (Beck depression score >21),
7. History of substance abuse or dependence within the past year, excluding nicotine and caffeine.
8. Serious or unstable cardiovascular, hepatic, renal, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical conditions (including unstable hypertension, hypo or hyperthyroidism, or psychological conditions that in the opinion of the investigators would compromise participation or be likely to lead to an adverse response, including injuries or hospitalization, during the course of the study. We will get the information from the health/activity questionnaire.
9. Have any DSM-IV Axis (major depression, addiction, anxiety) disorder which, in the judgment of the investigators, would interfere with compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Health/Activity Questionnaire | Baseline
The Fibromyalgia Impact Questionnaire | Baseline and end of 5th, 10th treatments and end of 1, 2, 3, 4, 5, and 6 months
Multidimensional Pain Inventory | Baseline and end of 5th, 10th treatments and end of 1, 2, 3, 4, 5, and 6 months
Beck Depression Inventory | Baseline and end of 5th, 10th treatments and end of 1, 2, 3, 4, 5, and 6 months

SECONDARY OUTCOMES:
30-sec Chair Stand | Baseline and end of 5th, 10th treatments and end of 1, 2, 3, 4, 5, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sivarama P Vinjamury, MD, MAOM, Principal Investigator — Southern California University of Health Sciences

REFERENCES:
- See also: Visit Southern California University of Health Sciences Website — http://www.scuhs.edu